CLINICAL TRIAL: NCT05187130
Title: The Effect of Mindfulnes Program on Stress, Depression and Psychological Well-being in Cancer Patients: Single Blinded Randomized Controlled Study
Brief Title: The Effect of Mindfulnes Program on Stress, Depression and Psychological Well-being in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant professor Dr., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Cancer patients mindfulness
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms; Cancer
Keywords: Stress, Psychological; Depression; Anxiety Disorders
MeSH Terms: conditions — Neoplasms; Stress, Psychological; Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mindfulness-based breathing and music therapy
  Interventions: Other: Mindfulness
- Control (No Intervention): No intervention has been made

INTERVENTIONS:
Other: Mindfulness — 60 patients in the mindfulness-based breathing and music therapy group were divided into subgroups of 5 participants each. Each 6-person group started by having participants complete the pretest State Anxiety Inventory, Beck Depression Inventory, and Psychological Well-Being Scale via Survey Monkey. Mindfulness-based breathing and music therapy was applied to each patient group in approximately 45-minute sessions per day. At the end of the session, participants re-filled the posttest State Anxiety Inventory, Work-Related Tension Scale, and Psychological Well-Being Scale. A total of 3 sessions were completed with an interval of two days.
  Arms: Intervention

SUMMARY:
Study design A single blinded, randomized controlled experimental design was used. The study complied with guidelines outlined under the Consolidated Standards of Reporting Trials (CONSORT) checklist.

Sample and Participants The study was carried out in July-December 2021 with the participation of cancer patients who were treated at a university hospital in Istanbul/Turkey.

Inclusion criteria; Patients aged 18 and over, volunteering to participate in the study, conscious and without communication problems, who did not take any course or practice (intervention?) on anxiety, tension, depression symptoms and coping with stress were included in the study. Participitants randomised intervention and controlled groups.

DETAILED DESCRIPTION:
Study design A single blinded, randomized controlled experimental design was used. The study complied with guidelines outlined under the Consolidated Standards of Reporting Trials (CONSORT) checklist.

Sample and Participants The study was carried out in July-December 2021 with the participation of cancer patients who were treated at a university hospital in Istanbul/Turkey.

Inclusion criteria; Patients aged 18 and over, volunteering to participate in the study, conscious and without communication problems, who did not take any course or intervention on anxiety, tension, depression symptoms and coping with stress were included in the study.

Sample size and randomization The sample number was calculated using the GPower 3.1.9 version program. At an effect size of 0.5 and an error level of 0.05 [alpha], the required sample size was determined to be at least 54 individuals for each group. A power analysis was performed considering the number of samples and the values of the data obtained from a similar study in the literature (Lee et al., 2020). The power of the analysis made with this sample size was determined as 93.1%. Considering the losses during the study, the sample number for each group was determined as 60 people.

The groups of participants who agreed to participate in the study were determined by the program with the randomization URL http://www.randomization.com/. In order to distribute the numbers to the groups, the numbers from 1 to 120 were randomly assigned to the two groups, assuming that set 1 would represent the intervention group and set 2 would represent the control group. In line with the program, the order of the patients forming the sample group was determined by randomization. A total of 130 patients, 65 in the intervention group and 65 in the control group, were included in the study. 5 participants in the intervention group who did not want to participate and died during the study, and 5 participants in the control group who did not want to participate and died during the study were not included in the evaluation. In the study, the results of a total of 120 patients, 60 in the intervention group and 60 in the control group, were analyzed.

Measures/Instruments Participant Information Form, State Anxiety Inventory, Beck Depression Inventory, and Psychological Well-Being Scale were used to collect research data. Survey Monkey was used as the data collection method. The Survey Monkey survey was created, which provides self-access and makes it easier to collect and track data by preventing multiple data entries from the same person. Confidentiality was ensured by completely disabling electronic and IP address registrations to receive anonymous responses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* volunteering to participate in the study,
* conscious and not having communication problems,
* not taking any course on anxiety, tension, depression symptoms and coping with stress

Exclusion Criteria:

* Diagnosed with a known psychiatric illness (delirium, anxiety, panic attack, depression) • Take another psychological relaxation course or training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Information Form | Baseline
  This form was developed by the researchers to include the age, gender, marital status, educational status, and treatment method of the participants.
State Anxiety Inventory | Baseline
  The State Anxiety Inventory was developed by Spielberger et al. in 1970 to determine the state anxiety levels of individuals. Turkish reliability and validity studies of the inventory were carried out by Öner and Le Compte (1983). The State Anxiety Inventory measures anxiety in adults. In the 20-item State Anxiety Inventory, the total score obtained from the four-point Likert-type inventory for each item can vary between 20 and 80. A high score indicates a high level of anxiety, while a small score indicates a low level of anxiety (Spielberger, et al., 1970; Öner & Le, 1983). Possible scores on the Scale range from 0 to 19 points (interpreted as meaning no state anxiety), 20 to 39 points (mild), 40 to 59 points (moderate), 60 to 79 points (severe), and 80 points and above ( very severe state anxiety).
State Anxiety Inventory | at the end of week 1
  The State Anxiety Inventory was developed by Spielberger et al. in 1970 to determine the state anxiety levels of individuals. Turkish reliability and validity studies of the inventory were carried out by Öner and Le Compte (1983). The State Anxiety Inventory measures anxiety in adults. In the 20-item State Anxiety Inventory, the total score obtained from the four-point Likert-type inventory for each item can vary between 20 and 80. A high score indicates a high level of anxiety, while a small score indicates a low level of anxiety (Spielberger, et al., 1970; Öner & Le, 1983). Possible scores on the Scale range from 0 to 19 points (interpreted as meaning no state anxiety), 20 to 39 points (mild), 40 to 59 points (moderate), 60 to 79 points (severe), and 80 points and above ( very severe state anxiety).
Psychological Well-Being Scale | baseline
  The scale, which was developed by Diener, Scollon, and Lucas, (2009) to measure the level of psychological well-being, has eight items. It identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life. The Turkish validity and reliability of the scale was made by Telef in 2013. Scale items are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). The Cronbach's alpha internal consistency coefficient of the scale was found to be 0.87. A high score from the scale indicates that the person has good psychological strength.
Psychological Well-Being Scale | at the end of week 1
  The scale, which was developed by Diener, Scollon, and Lucas, (2009) to measure the level of psychological well-being, has eight items. It identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life. The Turkish validity and reliability of the scale was made by Telef in 2013. Scale items are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). The Cronbach's alpha internal consistency coefficient of the scale was found to be 0.87. A high score from the scale indicates that the person has good psychological strength.
Beck Depression Inventory | baseline
  Beck et al. The validity and reliability study of the scale developed by Hisli in 1988 was carried out by Hisli. It is a depression rating scale consisting of 21 questions in total, evaluated by adding the scores between 0-3 obtained from each answer. Scale in line with the corresponding score intervals; 1-10 normal, 11-16 moderate mood disorder, 17-20 clinical depression; It is grouped as moderate depression between 21-30, severe depression between 31-40, and severe depression between 41-63.
Beck Depression Inventory | at the end of week 1.
  Beck et al. The validity and reliability study of the scale developed by Hisli in 1988 was carried out by Hisli. It is a depression rating scale consisting of 21 questions in total, evaluated by adding the scores between 0-3 obtained from each answer. Scale in line with the corresponding score intervals; 1-10 normal, 11-16 moderate mood disorder, 17-20 clinical depression; It is grouped as moderate depression between 21-30, severe depression between 31-40, and severe depression between 41-63.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek YILDIRIM, Ph.D, Study Director — Istanbul Aydın University
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)